CLINICAL TRIAL: NCT04275128
Title: Cooled Genicular Radiofrequency Ablation Versus Conventional Genicular Radiofrequency Ablation for the Treatment of Chronic Knee Pain: A Prospective Study
Brief Title: Cooled Versus Conventional Genicular Radiofrequency Ablation for Chronic Knee Pain
Status: Terminated | Type: Observational
Why Stopped: Insurance companies no longer cover this procedure
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Rohit Aiyer, Senior Staff Pain Medicine Physician, Henry Ford Health System
Other Study IDs: HFHSCooledRFAblation
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Chronic Knee Pain
Keywords: genicular ablation; cooled radiofrequency; chronic knee pain; cooled RF; radiofrequency ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Conventional Genicular Ablation: This group is scheduled to receive conventional genicular ablation to treat their chronic knee pain.
  Interventions: Device: Conventional radiofrequency ablation
- Cooled radiofrequency Ablation: This group is scheduled to receive cooled radiofrequency ablation to treat their chronic knee pain.
  Interventions: Device: Cooled radiofrequency ablation

INTERVENTIONS:
Device: Cooled radiofrequency ablation — Cooled radiofrequency thermal treatment uses the electrical current produced by radio waves to destroy a part of nerve tissue and relieve pain.
  Other Names: Cooled radiofrequency thermal treatment
  Groups: Cooled radiofrequency Ablation
Device: Conventional radiofrequency ablation — Genicular nerve ablation involves using radiofrequency to heat up the genicular nerve until it dies, causing relief of pain. This is a minimally invasive treatment that does not require any medication.
  Other Names: Genicular ablation; Genicular nerve ablation
  Groups: Conventional Genicular Ablation

SUMMARY:
This prospective observational study seeks to compare pain relief and disability following cooled radiofrequency ablation (Coolief) versus conventional genicular nerve ablation in patients with chronic knee pain. Patients' NRS for pain, WOMAC, and ODI score at baseline and 1, 3 and 6 months after treatment will be used to evaluate whether Coolief is more effective at reducing disability and improving pain relief.

DETAILED DESCRIPTION:
This prospective observational study seeks to compare pain relief at 1 month, 3 months and 6 months following cooled radiofrequency ablation vs conventional genicular nerve ablation in patients with chronic knee pain.

Both cooled RF and conventional genicular nerve ablation use the electrical current produced by radio waves to destroy a part of nerve tissue, creating a lesion and relieving pain (Kapural and Mekhail 2001). The conventional probe emanates heat that can damage surrounding tissues, and the lesion produced is limited in size. Cooled radiofrequency (RF) probes have a system of water running through the probe tip that keeps the probe tip at a lower temperature (Lorentzen 2015). Coolief produces larger spherical-shaped lesions, meaning an increased area of nerve destruction with less heat damage to surrounding tissues (Menzies and Hawkins 2015).

In 2017, the FDA cleared the Cooled radiofrequency thermal treatment device (Coolief, Halyard Health, Alpharetta, GA, USA) for knee osteoarthritis. McCormick et al investigated 33 patients with knee osteoarthritis pain, and after 6 months, 35% of patients had at least 50% or greater reduction in Numeric Rating Scale (NRS) for Pain, and 19% had complete pain relief. In another study by Davis et al, they compared, prospective, multicenter, randomized trial of 151 patients that compared cooled radiofrequency ablation genicular against intraarticular steroid injection. At 6 months, the cooled radiofrequency ablation group had more favorable outcomes in NRS: pain reduction 50% or greater was 74.1% in the ablation group versus 16.2% in the intraarticular group. Henry Ford Hospital Pain center introduced cooled radiofrequency ablation treatment modality in 2017 and it's currently being used in patients with chronic knee osteoarthritis and post-surgical knee pain.

This study will follow patients who have been diagnosed with chronic knee osteoarthritis or post-surgical knee pain and are scheduled to undergo Coolief or conventional ablation to treat their chronic knee pain. At 1, 3 and 6 months following their treatment, the study team will call patients on the phone to give them to ask about their pain and disability, using the NRS for pain, WOMAC for knee pain, and ODI questionnaire. Baseline and post-treatment scores will be compared to determine if Coolief elicits a more pronounced impact on reduced pain and disability than the conventional technique.

We expect to find a greater reduction in pain and disability experienced by patients who undergo the newer, cooled radiofrequency ablation when compared to the conventional ablation technique, at 1, 3- and 6-months after the procedure. The information gained from this study will be used to guide future ablation treatment, to ensure that patients receive the most effective pain relief treatment for their chronic knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (above age of 18)
* Diagnosed with chronic knee osteoarthritis or post Total Knee Arthroscopy or post Total Knee Replacement Pain
* More than 3 months of knee pain
* Scheduled for Genicular Knee ablation (Cooled or conventional ablation)
* Had previous intra articular injection (steroids or Hyaluronic acids) if not a post-surgical knee pain patient
* Achieved minimum 50% relief from genicular block x 2
* Numeric Rating Scale Score of 4 or greater
* Kellgren-Lawrence Knee Osteoarthritis Grade 2 or greater (in non post-surgical patients)

Exclusion Criteria:

* Pregnant adult female
* Patient fully anticoagulated
* Antiplatelet Use
* History of Clotting Disorder
* Refusal to participate
* Focal neurologic deficits
* Cognitive deficits
* History of Bone Cancer
* Mental Health Illness which causes instability
* Previous Knee radiofrequency ablation
* Active Infection
* Allergy to Medications Administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with chronic knee osteoarthritis or post-knee surgical pain, being treated with either cooled radiofrequency ablation at any of the five study locations (HFH Main and HFMC- Ford Rd, HFMC- Columbus, HFMC-Pierson, HFH West Bloomfield) between February 2020 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) Pain Score | 6 months
  This is a validated scale which consists of a rating of pain intensity from 0 (no pain) to 10 (worst possible pain). Score reported will be a number, and therefore a value between 0 to 10, with 0 meaning no pain to 10 meaning maximum pain (Krebs et al, 2007).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) knee pain score | 6 months
  The specific knee pain Short-form Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a validated questionnaire which measures pain, stiffness and functional limitation. Describe the details of the version you will be using. It is comprised of 24 items divided into three subscales: Pain (5 questions), stiffness (2 questions), and physical function (17 questions). Each question is scored on a scale of 0-4 with regards to severity, with 0 meaning no severity and 4 meaning extreme severity. Values are summed up for a combined WOMAC score, with 0 being the lowest, and 96 being the highest (or worst in severity with regards to pain, stiffness and limitations in function (Bellamy et al).
Oswestry Disability Index (ODI) | 6 months
  The Oswestry Disability Index (ODI) is a validated questionnaire used to quantify disability for low back pain. It consists of ten questions, each scored 0-5, with zero indicating the least amount of disability and 5 indicating the most severe disability. The scores are summed and multiplied by two to produce a final score ranging between 0 to 100, with zero meaning no disability and 100 meaning the maximum disability (Fairbank and Pynsent 2000).
Opioid dose after treatment | 1 day
  The opioid dose given to the patient after ablation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Aiyer, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapural L, Mekhail N. Radiofrequency ablation for chronic pain control. Curr Pain Headache Rep. 2001 Dec;5(6):517-25. doi: 10.1007/s11916-001-0069-z. PMID 11676886
- [Background] Lorentzen T. A cooled needle electrode for radiofrequency tissue ablation: thermodynamic aspects of improved performance compared with conventional needle design. Acad Radiol. 1996 Jul;3(7):556-63. doi: 10.1016/s1076-6332(96)80219-4. PMID 8796717
- [Background] Menzies RD, Hawkins JK. Analgesia and Improved Performance in a Patient Treated by Cooled Radiofrequency for Pain and Dysfunction Postbilateral Total Knee Replacement. Pain Pract. 2015 Jul;15(6):E54-8. doi: 10.1111/papr.12292. Epub 2015 Apr 10. PMID 25857719
- [Background] McCormick ZL, Korn M, Reddy R, Marcolina A, Dayanim D, Mattie R, Cushman D, Bhave M, McCarthy RJ, Khan D, Nagpal G, Walega DR. Cooled Radiofrequency Ablation of the Genicular Nerves for Chronic Pain due to Knee Osteoarthritis: Six-Month Outcomes. Pain Med. 2017 Sep 1;18(9):1631-1641. doi: 10.1093/pm/pnx069. PMID 28431129
- [Background] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley D, Patel N, Choi D, Soloman M, Gupta A, Desai M, Buvanendran A, Kapural L. Prospective, Multicenter, Randomized, Crossover Clinical Trial Comparing the Safety and Effectiveness of Cooled Radiofrequency Ablation With Corticosteroid Injection in the Management of Knee Pain From Osteoarthritis. Reg Anesth Pain Med. 2018 Jan;43(1):84-91. doi: 10.1097/AAP.0000000000000690. PMID 29095245